CLINICAL TRIAL: NCT02295722
Title: Infusional Gemcitabine and High-dose Melphalan (HDM) Conditioning Prior to (ASCT) Autologous Stem Cell Transplantation for Patients With Relapsed/Refractory Lymphoma
Brief Title: GEMHDM2014 : Gem-HDM HDT and ASCT for Relapsed/ Refractory Lymphoma
Acronym: GEMHDM2014
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: It did not show a significant benefit to justify completing the full target accrual.
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Tom Baker Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMHDM2014
Record Dates: First submitted 2014-10-30; First posted 2014-11-20 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Hodgkin's Lymphoma - Relapsed/Refractory; Non-Hodgkin's Lymphoma - Aggressive; Follicular Lymphoma
Keywords: eligible for high-dose therapy and stem cell transplantation
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Gemcitabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine/Melphalan Condition + ASCT (Experimental): Day -1 -
  * IV gemcitabine 1.5-2.5 g/m2 (depending on dose level assigned) administered as a loading bolus of 75 mg/m2, followed by a continuous infusion of 10 mg/m2/min.
  * immediately following gemcitabine - IV melphalan 200 mg/m2 over 5 minutes.
  Day 0
  •Stem cell infusion
  Patients will be assigned a dose level using the continual reassessment method based on the toxicity data available at the time of their enrollment. The dosing will start at 1.5 g/m2 and will increase by 0.5 mg/m2 at each level to a maximum of 2.5 g/m2. Dose-limiting toxicity is defined as grade 3 mucositis or skin toxicity lasting more than 3 days before downgrading, or any grade 4 non-hematological toxicity.
  Interventions: Drug: Gemcitabine; Drug: Melphalan; Other: ASCT

INTERVENTIONS:
Drug: Gemcitabine — gemcitabine 1.5 g/m2 INFUSED
Drug: Melphalan — 200 mg/m2
Other: ASCT — Day 0 - Stem cell infusion

SUMMARY:
Objective of study: To evaluate the safety and efficacy of infusional gemcitabine prior to HDM (high-dose melphalan) as HDCT (High Dose Chemotherapy) followed by autologous stem cell transplantation in patients with relapsed/refractory lymphoma.

DETAILED DESCRIPTION:
High-dose chemotherapy with autologous stem cell transplantation is the current standard of care for patients with chemosensitive relapsed Hodgkin's lymphoma and aggressive non-Hodgkin's lymphoma, and is an established effective therapy for patients with relapsed follicular lymphoma. Disease relapse remains a major problem, occurring in 50% of these patients, particularly in patients with primary refractory disease or other high-risk features. The addition of gemcitabine to single-agent melphalan as a high-dose conditioning regimen presents a promising combination that may lead to improvements in EFS (Event free survival). If this trial gives encouraging results, it may lead to a phase III trial evaluating this treatment strategy.

Drug exposure would be AUC (area under curve) and clinical factors would be things like obesity, renal function, disease characteristics.

We would be looking at the safety outcomes - i.e. adverse events as a measure of safety and tolerability. The adverse events would be non-hematological toxicities (any) and whether or not it is related to AUC. AUC in relationship to PFS (progression free survival) is also important (we want to know if we need to adjust dose to improve PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent
2. Age over 18 years
3. Relapsed/refractory lymphoma after at least 1 prior chemotherapy treatment:

   1. Hodgkin's lymphoma
   2. Aggressive non-Hodgkin's lymphoma
   3. Follicular lymphoma
4. Chemosensitive disease at time of transplantation (i.e. partial response or better to salvage chemotherapy)
5. ECOG (Eastern Cooperative Oncology Group) performance 0-2
6. Adequate organ function:

   1. Cardiac: LVEF (left ventricular ejection fraction)>40%
   2. Pulmonary: FEV1 (forced expiratory volume at one second) and DLCO (diffusing capacity of lung for carbon monoxide)>60% predicted
   3. Renal: creatinine <150 µmol/L unless caused by ureteric obstruction from lymphoma
   4. Liver: No evidence of cirrhosis. ALT (Alanine Aminotransferase) and bilirubin <2x upper limit of normal unless caused by biliary tract obstruction from lymphoma

Exclusion Criteria:

1. Clinically significant active infection
2. Active secondary central nervous system disease
3. Other serious co-morbid illness that would compromise study participation.
4. Pregnant or lactating females
5. Prior HDCT/ASCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04; Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Progression free survival of relapsed/refractory lymphoma patients treated with infusional gemcitabine, high dose melphalan (Gem-Mel) and ASCT | 3 years
  The goal is to improve overall 3-year PFS by 15% over what would be expected with standard conditioning regimens. Patients will be stratified into 3 groups according to disease: (a) relapsed/refractory Hodgkins's lymphoma, (b) relapsed/refractory aggressive non-Hodgkin's lymphoma, and (c) relapsed/refractory follicular lymphoma. Grade 3-4 non-hematological toxicity will be defined by the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.
Grade 3-4 Hematological Toxicity | 3 YEARS
  Assessment of Dose-limiting toxicity is defined as grade 3 mucositis or skin toxicity lasting more than 3 days before downgrading, or any grade 4 non-hematological toxicity.

SECONDARY OUTCOMES:
Overall survival | 3 Years
  The goal of this study is to improve overall 3-year PFS rate by 15% with the melphalan gemcitabine conditioning.
Cost Effectiveness | 3 Years
  Cost-effectiveness as measured by in-hospital costs of Gemcitabine-Melphalan relative to historical controls treated in Calgary with BEAM or Melphalan+/-TBI (Total Body Irradiation).
Measure of Melphalan pharmacokinetics, AUC (area under curve) | 3 Years
  Drug exposure would be AUC (area under curve) . Once the dose of gemcitabine has been established, all subsequent patients will receive a uniform HDCT (high dose chemotherapy) regimen. Patients will undergo blood draws for pharmacokinetic testing at the following time points relative to the end of melphalan infusion: 5 minutes, 30 minutes, 1 hour, 3 hours, 5 hours, 7-10 hours, and 18-23 hours. Samples will be processed at the local pharmacokinetics laboratory in Calgary
Evaluation of relationship between clinical factors and drug exposure in treatment of Gemcitabine/Melphalan with ASCT (autologous stem cell transplantation) | 3 years
  The number of patients with adverse events as a measure of safety and tolerability.
Evaluation of relation between drug exposure and non-hematological toxicity and progression free survival | 3 years
  Drug exposure as measured by area under the curve related to number of patients with adverse events (non-hematological toxicity) and progression-free survival
Safety Outcomes assessed adverse events as a measure of safety and tolerability | 3 years
  Assess adverse events as a measure of safety and tolerability. The adverse events would be non-hematological toxicities (any) and whether or not it is related to AUC. AUC in relationship to PFS is also important (we want to know if we need to adjust dose to improve PFS).

CONTACTS AND LOCATIONS:
Overall Officials: MONA SHAFEY, MD, Principal Investigator — Tom Baker Cancer Centre
Locations (1):
- Tom Baker Cancer Center, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No